CLINICAL TRIAL: NCT03208010
Title: Diabetes Prevention Culturally Tailored for Mexican Americans
Brief Title: Diabetes Prevention for Mexican Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sharon A Brown, PhD, Professor Emeritus and Senior Research Scientist, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DK109920 (NIH)
Record Dates: First submitted 2017-06-22; First posted 2017-07-05 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Prediabetic State; Overweight and Obesity
Keywords: health disparities; lifestyle behaviors; diabetes prevention; Hispanic health
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The study involves an examination of the effectiveness of a culturally-tailored diabetes prevention intervention using a randomized, repeated measures, pretest/post-test control group design. Groups are randomly assigned to: 1) the diabetes prevention intervention; or 2) an "enhanced" usual care control group. Outcome measurements are made at 3, 6, 12, 24, and 36 months post entry into the study to examine changes over time in key diabetes and health indicators.
Masking Description: Given the nature of behavioral programs, we are not able to mask participant involvement. Some primary care providers may not know the details of their patients' participation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Intervention (Experimental): The intervention is 12 weeks of education on diet and physical activity, followed by 15 biweekly support groups for problem solving. Then, 3 booster sessions are scheduled, each one at 6-month intervals. Further, motivational interviewing is infused into all group sessions.
  Interventions: Behavioral: Diabetes Prevention Intervention
- Enhanced Usual Care (Active Comparator): The comparator is an "enhanced" usual care control group that receives health care from personal physicians plus has access to: a) data collection sessions; b) individualized exit interviews with program staff after each data collection session to receive immediate feedback on lab results and trends in personal health indicators (e.g., BMI, A1C) and to ask questions; c) referral to a local physician or clinic, if needed; and d) Spanish-language materials on diabetes prevention.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Diabetes Prevention Intervention — * Educational sessions with emphasis on physical activity, healthy cultural diets, and strategies to promote positive behavioral changes.
  * Specific goals set for weight loss and physical activities
  * Fitbits provided for monitoring physical activity goals
  * Weekly review of and feedback on effects of physical activity (Fitbits) and dietary changes (checklists)
  * 15 biweekly support group sessions plus 3 booster sessions every 6 months thereafter
  Note: In response to the COVID-19 pandemic, a remote version of the intervention was designed to provide the program remotely instead of via the usual in-person group format. This alternative strategy is designed to replace the biweekly support groups, which in the past focused on similar content, i.e., reviewing key educational content, demonstrations of healthy Mexican American recipes.
  Other Names: Culturally Tailored Diabetes Prevention
  Arms: Diabetes Prevention Intervention
Other: Enhanced Usual Care — * Monitoring by existing personal physicians
  * Feedback on lab results
  * Referrals to physicians or clinics, if needed
  * Diabetes prevention educational materials
  Arms: Enhanced Usual Care

SUMMARY:
This study tests a culturally tailored lifestyle intervention designed to prevent, or delay onset of, T2DM in Mexican Americans with prediabetes. Half the participants take part in a lifestyle program that emphasizes preparing and eating healthy Mexican American foods and increasing physical activity; the other half take part in an "enhanced" usual care control group.

DETAILED DESCRIPTION:
The main purpose of this study is to test a culturally tailored lifestyle intervention that incorporates motivational interviewing and is designed to prevent, or delay onset of, T2DM in Mexican Americans with prediabetes. Groups of participants are randomly assigned to: a) an experimental group that receives a lifestyle program (12 2-hour weekly educational group sessions) that emphasizes preparing and eating healthy Mexican American foods and increasing physical activity, followed by 14 biweekly support group sessions to problem solve remaining barriers to adopting recommended behaviors and 3 booster sessions to enhance maintenance of behavioral changes; OR b) an "enhanced" usual care control group that receives lab results with individualized guidance and referrals. A secondary goal of the study is to examine the influence of genetic variation at selected candidate genes for glucose regulation on response to the lifestyle intervention.

The specific aims of the study are to:

1. Test a culturally tailored lifestyle intervention that incorporates motivational interviewing and is designed to prevent, or delay onset of, T2DM in Mexican Americans with prediabetes. Groups of participants are randomly assigned to: a) an experimental group that receives a lifestyle program (12 2-hour weekly educational group sessions) that emphasizes preparing and eating healthy Mexican American foods and increasing physical activity, followed by 14 biweekly support group sessions to problem solve remaining barriers to adopting recommended behaviors and 3 booster sessions to enhance maintenance of behavioral changes; OR b) an "enhanced" usual care control group that receives lab results with individualized guidance and referrals.

   H1: The experimental group, compared to the control group, will have better health outcomes at 3, 6, 12, 24, and 36 months post baseline: 2-hour OGTT, A1C, FBG, lipids, blood pressure, health behaviors (physical activity, dietary intake), health beliefs: barriers, and anthropometrics (BMI [primary outcome], waist circumference). Other baseline measures - demographics and acculturation - characterize the population and correct for any baseline imbalances between groups.
2. Prior to testing the intervention, we conduct focus groups in Starr County with participants of our previous DSMES studies, physicians from both sides of the border, local health officials, and key authority figures (Catholic priests, county officials) to fine tune intervention aspects in the context of diabetes prevention.
3. Exploratory Aim: Examine the influence of genetic variation at selected candidate genes for glucose regulation on response to the lifestyle intervention.

The study addresses THE major public health problem of U.S.-Mexico border communities.

Note: In response to the COVID-19 pandemic, a remote version of the intervention was designed to provide the program remotely instead of via the usual in-person group format. A series of augmented text messages were developed that included 5 to 10-minute videos of a project dietitian or nurse talking about previously-learned content and demonstrating a simple, healthier method of preparing favorite recipe(s). The URLs of other related Spanish-language videos from the Internet are included and the text messages with videos are supplemented with phone calls from community workers to provide follow-up coaching for motivation. This alternative strategy is designed to replace the biweekly support groups, which in the past focused on similar content, i.e., reviewing key educational content, demonstrations of healthy Mexican American recipes.

ELIGIBILITY:
Inclusion Criteria:

* no prior diabetes diagnosis (except gestational)
* impaired fasting glucose (fasting glucose between 100 and 125 mg/dL) OR impaired glucose tolerance (between 140 and 199 mg/dL on a 2-hour post-load glucose tolerance test) OR A1C between 5.7% and 6.4%)
* have not previously participated in diabetes self-management education studies
* Mexican American

Exclusion Criteria:

* diagnosed with diabetes at baseline
* fasting glucose greater than or equal to 126 mg/dL
* ever used hypoglycemic medication (except during pregnancy)
* are currently pregnant or within 3 months postpartum
* are migrant farmworkers who migrate for more than 2 weeks
* take medications that could confound a diabetes diagnosis (e.g., steroids)
* have medical conditions for which changes in diet and/or physical activity would be contraindicated

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin (A1C) at 3 months | Baseline and 3 months
  A1C, an indicator of long-term glucose control, is measured as the percentage of red blood cells that are glycosylated (have a glucose molecule connected) and is analyzed onsite using a point-of-care device (Siemens DCA Vantage Analyzer, Malvern, PA).
Change from baseline in glycosylated hemoglobin (A1C) at 6 months | Baseline and 6 months
  A1C, an indicator of long-term glucose control, is measured as the percentage of red blood cells that are glycosylated (have a glucose molecule connected) and is analyzed onsite using a point-of-care device (Siemens DCA Vantage Analyzer, Malvern, PA).
Change from baseline in glycosylated hemoglobin (A1C) at 12 months | Baseline and 12 months
  A1C, an indicator of long-term glucose control, is measured as the percentage of red blood cells that are glycosylated (have a glucose molecule connected) and is analyzed onsite using a point-of-care device (Siemens DCA Vantage Analyzer, Malvern, PA).
Change from baseline in glycosylated hemoglobin (A1C) at 24 months | Baseline and 24 months
  A1C, an indicator of long-term glucose control, is measured as the percentage of red blood cells that are glycosylated (have a glucose molecule connected) and is analyzed onsite using a point-of-care device (Siemens DCA Vantage Analyzer, Malvern, PA).
Change from baseline in glycosylated hemoglobin (A1C) at 36 months | Baseline and 36 months
  A1C, an indicator of long-term glucose control, is measured as the percentage of red blood cells that are glycosylated (have a glucose molecule connected) and is analyzed onsite using a point-of-care device (Siemens DCA Vantage Analyzer, Malvern, PA).
Change from baseline in body mass index (BMI) at 3 months | Baseline and 3 months
  Body weights are measured with a balance beam scale with individuals in street clothing and without shoes. Heights are obtained using a secured stadiometer. BMI is calculated (weight(kg)/height/meters^2).
Change from baseline in body mass index (BMI) at 6 months | Baseline and 6 months
  Body weights are measured with a balance beam scale with individuals in street clothing and without shoes. Heights are obtained using a secured stadiometer. BMI is calculated (weight(kg)/height/meters^2).
Change from baseline in body mass index (BMI) at 12 months | Baseline and 12 months
  Body weights are measured with a balance beam scale with individuals in street clothing and without shoes. Heights are obtained using a secured stadiometer. BMI is calculated (weight(kg)/height/meters^2).
Change from baseline in body mass index (BMI) at 24 months | Baseline and 24 months
  Body weights are measured with a balance beam scale with individuals in street clothing and without shoes. Heights are obtained using a secured stadiometer. BMI is calculated (weight(kg)/height/meters^2).
Change from baseline in body mass index (BMI) at 36 months | Baseline and 36 months
  Body weights are measured with a balance beam scale with individuals in street clothing and without shoes. Heights are obtained using a secured stadiometer. BMI is calculated (weight(kg)/height/meters^2).

SECONDARY OUTCOMES:
Change from baseline to 3 months in quality of life as measured with 1 researcher-developed item | Baseline and 3 months
  Measured with 1 item developed by the research team. The participants respond to the following statement -- "In general, my well being is..." Item responses range from 1-7, with 7 indicating as good as it possibly could be and 1 indicating as bad as it possibly could be. The item employs a 1-7 Likert-type scale with higher numbers indicating a more favorable perceived quality of life.
Change from baseline to 12 months in quality of life as measured with 1 researcher-developed item | Baseline and 12 months
  Measured with 1 item developed by the research team. The participants respond to the following statement -- "In general, my well being is..." Item responses range from 1-7, with 7 indicating as good as it possibly could be and 1 indicating as bad as it possibly could be. The item employs a 1-7 Likert-type scale with higher numbers indicating a more favorable perceived quality of life.
Change from baseline to 24 months in quality of life as measured with 1 researcher-developed item | Baseline and 24 months
  Measured with 1 item developed by the research team. The participants respond to the following statement -- "In general, my well being is..." Item responses range from 1-7, with 7 indicating as good as it possibly could be and 1 indicating as bad as it possibly could be. The item employs a 1-7 Likert-type scale with higher numbers indicating a more favorable perceived quality of life.
Change from baseline to 36 months in quality of life as measured with 1 researcher-developed item | Baseline and 36 months
  Measured with 1 item developed by the research team. The participants respond to the following statement -- "In general, my well being is..." Item responses range from 1-7, with 7 indicating as good as it possibly could be and 1 indicating as bad as it possibly could be. The item employs a 1-7 Likert-type scale with higher numbers indicating a more favorable perceived quality of life.
Changes from baseline to 12 months in number/amount of times foods were eaten during the previous month using the questionnaire entitled, Food Frequency Questionnaire for Starr County Health Studies (see McPherson et al., Ann Epidemiol, 1995). | Baseline and 12 months
  The Food Frequency Questionnaire for Starr County Studies lists 106 specific food items. The participants indicate the frequency a specific food item, including cultural foods, was eaten during the past month, as well as the portion size. For example, for the item "Cheetos," the respondent answers "yes" or "no" regarding whether the item was eaten during the past month. If "yes," then the individual is asked how many times and then asked to estimate portion size using food models available during the administration of the questionnaire. Special software enables converting frequency data to raw intake as well as nutrient densities for analysis. Macro- and micro-nutrients that will be quantified are: total caloric intake, protein, fat, saturated fat, mono-unsaturated fat, poly-unsaturated fat, cholesterol, carbohydrate intake, vitamins A, and E, carotene, calcium, and iron.
Changes from baseline to 24 months in number/amount of times foods were eaten during the previous month using the questionnaire entitled, Food Frequency Questionnaire for Starr County Health Studies (see McPherson et al., Ann Epidemiol, 1995) | Baseline and 24 months
  The Food Frequency Questionnaire for Starr County Studies lists 106 specific food items. The participants indicate the frequency a specific food item, including cultural foods, was eaten during the past month, as well as the portion size. For example, for the item "Cheetos," the respondent answers "yes" or "no" regarding whether the item was eaten during the past month. If "yes," then the individual is asked how many times and then asked to estimate portion size using food models available during the administration of the questionnaire. Special software enables converting frequency data to raw intake as well as nutrient densities for analysis. Macro- and micro-nutrients that will be quantified are: total caloric intake, protein, fat, saturated fat, mono-unsaturated fat, poly-unsaturated fat, cholesterol, carbohydrate intake, vitamins A, and E, carotene, calcium, and iron.
Changes from baseline to 36 months in number/amount of times foods were eaten during the previous month using the questionnaire entitled, Food Frequency Questionnaire for Starr County Health Studies (see McPherson et al., Ann Epidemiol, 1995) | Baseline and 36 months
  The Food Frequency Questionnaire for Starr County Studies lists 106 specific food items. The participants indicate the frequency a specific food item, including cultural foods, was eaten during the past month, as well as the portion size. For example, for the item "Cheetos," the respondent answers "yes" or "no" regarding whether the item was eaten during the past month. If "yes," then the individual is asked how many times and then asked to estimate portion size using food models available during the administration of the questionnaire. Special software enables converting frequency data to raw intake as well as nutrient densities for analysis. Macro- and micro-nutrients that will be quantified are: total caloric intake, protein, fat, saturated fat, mono-unsaturated fat, poly-unsaturated fat, cholesterol, carbohydrate intake, vitamins A, and E, carotene, calcium, and iron.
Changes from baseline to 3 months in the number of times high-fat foods were eaten during the previous month using the Saturated Fat/Cholesterol Avoidance Scale, a culturally-tailored instrument developed in Starr County | Baseline and 3 months
  The Saturated Fat/Cholesterol Avoidance Scale is a brief 7-item scale that collects information on intake and use of saturated fat in the diet during the previous month. A major emphasis in the diet instruction is how to reduce lard when preparing Mexican-American recipes. Questions on the Scale are specific to Mexican-American foods, e.g., "When you eat refried beans, what type of fat are they made with?" The Scale is a brief 7-item scale and item responses range from 1 to 4, representing never to always. Higher scores reflect higher intake of high-fat foods.
Changes from baseline to 6 months in the number of times high-fat foods were eaten during the previous month using the Saturated Fat/Cholesterol Avoidance Scale, a culturally-tailored instrument developed in Starr County | Baseline and 6 months
  The Saturated Fat/Cholesterol Avoidance Scale is a brief 7-item scale that collects information on intake and use of saturated fat in the diet during the previous month. A major emphasis in the diet instruction is how to reduce lard when preparing Mexican-American recipes. Questions on the Scale are specific to Mexican-American foods, e.g., "When you eat refried beans, what type of fat are they made with?" The Scale is a brief 7-item scale and item responses range from 1 to 4, representing never to always. Higher scores reflect higher intake of high-fat foods.
Changes from baseline to 12 months in the number of times high-fat foods were eaten during the previous month using the Saturated Fat/Cholesterol Avoidance Scale, a culturally-tailored instrument developed in Starr County | Baseline and 12 months
  The Saturated Fat/Cholesterol Avoidance Scale is a brief 7-item scale that collects information on intake and use of saturated fat in the diet during the previous month. A major emphasis in the diet instruction is how to reduce lard when preparing Mexican-American recipes. Questions on the Scale are specific to Mexican-American foods, e.g., "When you eat refried beans, what type of fat are they made with?" The Scale is a brief 7-item scale and item responses range from 1 to 4, representing never to always. Higher scores reflect higher intake of high-fat foods.
Changes from baseline to 24 months in the number of times high-fat foods were eaten during the previous month using the Saturated Fat/Cholesterol Avoidance Scale, a culturally-tailored instrument developed in Starr County | Baseline and 24 months
  The Saturated Fat/Cholesterol Avoidance Scale is a brief 7-item scale that collects information on intake and use of saturated fat in the diet during the previous month. A major emphasis in the diet instruction is how to reduce lard when preparing Mexican-American recipes. Questions on the Scale are specific to Mexican-American foods, e.g., "When you eat refried beans, what type of fat are they made with?" The Scale is a brief 7-item scale and item responses range from 1 to 4, representing never to always. Higher scores reflect higher intake of high-fat foods.
Changes from baseline to 36 months in the number of times high-fat foods were eaten during the previous month using the Saturated Fat/Cholesterol Avoidance Scale, a culturally-tailored instrument developed in Starr County | Baseline and 36 months
  The Saturated Fat/Cholesterol Avoidance Scale is a brief 7-item scale that collects information on intake and use of saturated fat in the diet during the previous month. A major emphasis in the diet instruction is how to reduce lard when preparing Mexican-American recipes. Questions on the Scale are specific to Mexican-American foods, e.g., "When you eat refried beans, what type of fat are they made with?" The Scale is a brief 7-item scale and item responses range from 1 to 4, representing never to always. Higher scores reflect higher intake of high-fat foods.
Change from baseline to 3 months in weekly average of daily steps walked using a Fitbit activity tracker | Baseline and 3 months
  Each participant in the experimental group receives a free Fitbit activity tracker to monitor daily steps. An individual walking prescription is negotiated with each participant, with the general goal of individuals walking 10,000 steps per day. Walking data are automatically downloaded into secured software (Fitabase) for tracking.
Change from baseline to 6 months in weekly average of daily steps walked using a Fitbit activity tracker | Baseline and 6 months
  Each participant in the experimental group receives a free Fitbit activity tracker to monitor daily steps. An individual walking prescription is negotiated with each participant, with the general goal of individuals walking 10,000 steps per day. Walking data are automatically downloaded into secured software (Fitabase) for tracking.
Change from baseline to 12 months in weekly average of daily steps walked using a Fitbit activity tracker | Baseline and 12 months
  Each participant in the experimental group receives a free Fitbit activity tracker to monitor daily steps. An individual walking prescription is negotiated with each participant, with the general goal of individuals walking 10,000 steps per day. Walking data are automatically downloaded into secured software (Fitabase) for tracking.
Change from baseline to 24 months in weekly average of daily steps walked using a Fitbit activity tracker | Baseline and 24 months
  Each participant in the experimental group receives a free Fitbit activity tracker to monitor daily steps. An individual walking prescription is negotiated with each participant, with the general goal of individuals walking 10,000 steps per day. Walking data are automatically downloaded into secured software (Fitabase) for tracking.
Change from baseline to 36 months in weekly average of daily steps walked using a Fitbit activity tracker | Baseline and 36 months
  Each participant in the experimental group receives a free Fitbit activity tracker to monitor daily steps. An individual walking prescription is negotiated with each participant, with the general goal of individuals walking 10,000 steps per day. Walking data are automatically downloaded into secured software (Fitabase) for tracking.
Change from baseline to 3 months in perceived barriers to improving dietary habits using the Givens & Givens health beliefs: barriers subscale adapted for Starr County studies | Baseline and 3 months
  The Health Beliefs: Barriers questionnaire is a subscale from the health belief instrument adapted from the Givens & Givens Health Belief Scale. The instrument focuses on the barriers to following a prescribed diet. The instrument is a 12-item questionnaire and involves a Likert-type scale of 1-5; total scores range from 12 to 60 with higher scores indicating more barriers.
Change from baseline to 6 months in perceived barriers to improving dietary habits using the Givens & Givens health beliefs: barriers subscale adapted for Starr County studies | Baseline and 6 months
  The Health Beliefs: Barriers questionnaire is a subscale from the health belief instrument adapted from the Givens & Givens Health Belief Scale. The instrument focuses on the barriers to following a prescribed diet. The instrument is a 12-item questionnaire and involves a Likert-type scale of 1-5; total scores range from 12 to 60 with higher scores indicating more barriers.
Change from baseline to 12 months in perceived barriers to improving dietary habits using the Givens & Givens health beliefs: barriers subscale adapted for Starr County studies | Baseline and 12 months
  The Health Beliefs: Barriers questionnaire is a subscale from the health belief instrument adapted from the Givens & Givens Health Belief Scale. The instrument focuses on the barriers to following a prescribed diet. The instrument is a 12-item questionnaire and involves a Likert-type scale of 1-5; total scores range from 12 to 60 with higher scores indicating more barriers.
Change from baseline to 24 months in perceived barriers to improving dietary habits using the Givens & Givens health beliefs: barriers subscale adapted for Starr County studies | Baseline and 24 months
  The Health Beliefs: Barriers questionnaire is a subscale from the health belief instrument adapted from the Givens & Givens Health Belief Scale. The instrument focuses on the barriers to following a prescribed diet. The instrument is a 12-item questionnaire and involves a Likert-type scale of 1-5; total scores range from 12 to 60 with higher scores indicating more barriers.
Change from baseline to 36 months in perceived barriers to improving dietary habits using the Givens & Givens health beliefs: barriers subscale adapted for Starr County studies | Baseline and 36 months
  The Health Beliefs: Barriers questionnaire is a subscale from the health belief instrument adapted from the Givens & Givens Health Belief Scale. The instrument focuses on the barriers to following a prescribed diet. The instrument is a 12-item questionnaire and involves a Likert-type scale of 1-5; total scores range from 12 to 60 with higher scores indicating more barriers.
Change from baseline in blood cholesterol levels at 12 months | Baseline and 12 months
  Standard procedures for measuring cholesterol include the use of the Monotest Cholesterol procedure. The test is adapted to automatic analysis using the Hitachi 911 analyzer, a totally self-contained computerized, programmable, fully automated chemistry analyzer.
Change from baseline in blood cholesterol levels at 24 months | Baseline and 24 months
  Standard procedures for measuring cholesterol include the use of the Monotest Cholesterol procedure. The test is adapted to automatic analysis using the Hitachi 911 analyzer, a totally self-contained computerized, programmable, fully automated chemistry analyzer.
Change from baseline in blood cholesterol levels at 36 months | Baseline and 36 months
  Standard procedures for measuring cholesterol include the use of the Monotest Cholesterol procedure. The test is adapted to automatic analysis using the Hitachi 911 analyzer, a totally self-contained computerized, programmable, fully automated chemistry analyzer.
Change from baseline in blood triglyceride levels at 12 months | Baseline and 12 months
  Standard procedures for measuring triglycerides include the GPO Triglyceride procedure of Boehringer Mannheim. The test is adapted to automatic analysis using the Hitachi 911 analyzer. The Hitachi 911 analyzer is a totally self-contained computerized, programmable, fully automated chemistry analyzer.
Change from baseline in blood triglyceride levels at 24 months | Baseline and 24 months
  Standard procedures for measuring triglycerides include the GPO Triglyceride procedure of Boehringer Mannheim. The test is adapted to automatic analysis using the Hitachi 911 analyzer. The Hitachi 911 analyzer is a totally self-contained computerized, programmable, fully automated chemistry analyzer.
Change from baseline in blood triglyceride levels at 36 months | Baseline and 36 months
  Standard procedures for measuring triglycerides include the GPO Triglyceride procedure of Boehringer Mannheim. The test is adapted to automatic analysis using the Hitachi 911 analyzer. The Hitachi 911 analyzer is a totally self-contained computerized, programmable, fully automated chemistry analyzer.
Change from baseline in 2 hr.-Oral Glucose Tolerance Test (OGTT) at 12 months | Baseline and 12 months
  A simplified 2-hour OGTT is used with blood collection while fasting and 120 minutes following a 75-gram liquid glucose challenge. These procedures enable classification of prediabetes and diabetes according to all current recommendations.
Change from baseline in 2 hr.-Oral Glucose Tolerance Test (OGTT) at 24 months | Baseline and 24 months
  A simplified 2-hour OGTT is used with blood collection while fasting and 120 minutes following a 75-gram liquid glucose challenge. These procedures enable classification of prediabetes and diabetes according to all current recommendations.
Change from baseline in 2 hr.-Oral Glucose Tolerance Test (OGTT) at 36 months | Baseline and 36 months
  A simplified 2-hour OGTT is used with blood collection while fasting and 120 minutes following a 75-gram liquid glucose challenge. These procedures enable classification of prediabetes and diabetes according to all current recommendations.
Change from baseline in blood pressure at 3 months | Baseline and 3 months
  Blood pressure readings are taken using an automated device (Critikon Dinamap, Tampa, FL) following 5 minutes of sitting quietly. Measures of systolic (SBP) and diastolic (DBP) blood pressures involve averaging the second and third measures.
Change from baseline in blood pressure at 6 months | Baseline and 6 months
  Blood pressure readings are taken using an automated device (Critikon Dinamap, Tampa, FL) following 5 minutes of sitting quietly. Measures of systolic (SBP) and diastolic (DBP) blood pressures involve averaging the second and third measures.
Change from baseline in blood pressure at 12 months | Baseline and 12 months
  Blood pressure readings are taken using an automated device (Critikon Dinamap, Tampa, FL) following 5 minutes of sitting quietly. Measures of systolic (SBP) and diastolic (DBP) blood pressures involve averaging the second and third measures.
Change from baseline in blood pressure at 24 months | Baseline and 24 months
  Blood pressure readings are taken using an automated device (Critikon Dinamap, Tampa, FL) following 5 minutes of sitting quietly. Measures of systolic (SBP) and diastolic (DBP) blood pressures involve averaging the second and third measures.
Change from baseline in blood pressure at 36 months | Baseline and 36 months
  Blood pressure readings are taken using an automated device (Critikon Dinamap, Tampa, FL) following 5 minutes of sitting quietly. Measures of systolic (SBP) and diastolic (DBP) blood pressures involve averaging the second and third measures.
Change from baseline in depression measured with the Patient Health Questionnaire (PHQ-9) at 3 months | Baseline and 3 months
  The Patient Health Questionnaire (PHQ-9) is a brief, 9-item instrument to screen for depression. It employs a 0 to 3 scale: not at all, several days, more than half the days, and nearly every day. A composite score of 5-9 indicates mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-17 severe depression.
Change from baseline in depression measured with the Patient Health Questionnaire (PHQ-9) at 6 months | Baseline and 6 months
  The Patient Health Questionnaire (PHQ-9) is a brief, 9-item instrument to screen for depression. It employs a 0 to 3 scale: not at all, several days, more than half the days, and nearly every day. A composite score of 5-9 indicates mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-17 severe depression.
Change from baseline in depression measured with the Patient Health Questionnaire (PHQ-9) at 12 months | Baseline and 12 months
  The Patient Health Questionnaire (PHQ-9) is a brief, 9-item instrument to screen for depression. It employs a 0 to 3 scale: not at all, several days, more than half the days, and nearly every day. A composite score of 5-9 indicates mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-17 severe depression.
Change from baseline in depression measured with the Patient Health Questionnaire (PHQ-9) at 24 months | Baseline and 24 months
  The Patient Health Questionnaire (PHQ-9) is a brief, 9-item instrument to screen for depression. It employs a 0 to 3 scale: not at all, several days, more than half the days, and nearly every day. A composite score of 5-9 indicates mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-17 severe depression.
Change from baseline in depression measured with the Patient Health Questionnaire (PHQ-9) at 36 months | Baseline and 36 months
  The Patient Health Questionnaire (PHQ-9) is a brief, 9-item instrument to screen for depression. It employs a 0 to 3 scale: not at all, several days, more than half the days, and nearly every day. A composite score of 5-9 indicates mild depression; 10-14 moderate depression; 15-19 moderately severe depression; and 20-17 severe depression.
Change from baseline in confidence to improve dietary behaviors, using the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF) at 3 months | Baseline and 3 months
  The Weight Efficacy Lifestyle Questionnaire, an 8-item instrument, measures how confident (or certain) one is that he/she will be able to resist overeating in a number of difficult situations, such as in social settings or watching TV. The scale is a Likert-type scale of 0 (not confident) to 10 (very confident). Total scores range from 0-80 and higher scores indicate higher self-efficacy.
Change from baseline in confidence to improve dietary behaviors, using the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF) at 6 months | Baseline and 6 months
  The Weight Efficacy Lifestyle Questionnaire, an 8-item instrument, measures how confident (or certain) one is that he/she will be able to resist overeating in a number of difficult situations, such as in social settings or watching TV. The scale is a Likert-type scale of 0 (not confident) to 10 (very confident). Total scores range from 0-80 and higher scores indicate higher self-efficacy.
Change from baseline in confidence to improve dietary behaviors, using the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF) at 12 months | Baseline and 12 months
  The Weight Efficacy Lifestyle Questionnaire, an 8-item instrument, measures how confident (or certain) one is that he/she will be able to resist overeating in a number of difficult situations, such as in social settings or watching TV. The scale is a Likert-type scale of 0 (not confident) to 10 (very confident). Total scores range from 0-80 and higher scores indicate higher self-efficacy.
Change from baseline in confidence to improve dietary behaviors, using the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF) at 24 months | Baseline and 24 months
  The Weight Efficacy Lifestyle Questionnaire, an 8-item instrument, measures how confident (or certain) one is that he/she will be able to resist overeating in a number of difficult situations, such as in social settings or watching TV. The scale is a Likert-type scale of 0 (not confident) to 10 (very confident). Total scores range from 0-80 and higher scores indicate higher self-efficacy.
Change from baseline in confidence to improve dietary behaviors, using the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF) at 36 months | Baseline and 36 months
  The Weight Efficacy Lifestyle Questionnaire, an 8-item instrument, measures how confident (or certain) one is that he/she will be able to resist overeating in a number of difficult situations, such as in social settings or watching TV. The scale is a Likert-type scale of 0 (not confident) to 10 (very confident). Total scores range from 0-80 and higher scores indicate higher self-efficacy.
Change from baseline in perceived stress at 12 months | Change from baseline to 12 months
  To measure perceived stress, the NIH PROMIS questionnaire on perceived stress was added to the data collection plan. The instrument is a 10-item scale and each item is rated as 1 (never) to 5 (very often). Total scores range from 10 to 50, with higher scores indicating higher levels of perceived stress.
Change from baseline in perceived stress at 24 months | Change from baseline to 24 months
  To measure perceived stress, the NIH PROMIS questionnaire on perceived stress was added to the data collection plan. The instrument is a 10-item scale and each item is rated as 1 (never) to 5 (very often). Total scores range from 10 to 50, with higher scores indicating higher levels of perceived stress.
Change from baseline in perceived stress at 36 months | Change from baseline to 36 months
  To measure perceived stress, the NIH PROMIS questionnaire on perceived stress was added to the data collection plan. The instrument is a 10-item scale and each item is rated as 1 (never) to 5 (very often). Total scores range from 10 to 50, with higher scores indicating higher levels of perceived stress.
Text Messages Intervention - Follow-up Phone Call Interview | 1 week after distribution of the videos
  To measure participant satisfaction with the augmented text messaging revision to the intervention (in response to COVID-19 restrictions), the investigators developed a brief guide for follow-up phone interviews. Five questions are asked regarding changes in health, messages they remember from the video(s), questions they may have, preferences (text messages vs. in-person group sessions), and willingness to continue receiving future text messages.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Brown, PhD, Principal Investigator — University of Texas at Austin; Craig L. Hanis, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Starr County Research Field Office, Rio Grande City, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown SA, Perkison WB, Garcia AA, Cuevas HE, Velasquez MM, Winter MA, Hanis CL. The Starr County Border Health Initiative: Focus Groups on Diabetes Prevention in Mexican Americans. Diabetes Educ. 2018 Jun;44(3):293-306. doi: 10.1177/0145721718770143. Epub 2018 Apr 12. PMID 29644932
- [Result] Essigmann HT, Aguilar DA, Perkison WB, Bay KG, Deaton MR, Brown SA, Hanis CL, Brown EL. Epidemiology of Antibiotic Use and Drivers of Cross-Border Procurement in a Mexican American Border Community. Front Public Health. 2022 Mar 10;10:832266. doi: 10.3389/fpubh.2022.832266. eCollection 2022. PMID 35356027
- [Result] Brown SA, Becker HA, Garcia AA, Velasquez MM, Tanaka H, Winter MA, Perkison WB, Brown EL, Aguilar D, Hanis CL. The effects of gender and country of origin on acculturation, psychological factors, lifestyle factors, and diabetes-related physiological outcomes among Mexican Americans: The Starr County diabetes prevention initiative. Chronic Illn. 2023 Jun;19(2):444-457. doi: 10.1177/17423953221089315. Epub 2022 Mar 24. PMID 35331025
- [Result] Brown SA, Becker HA, Garcia AA, Velasquez MM, Tanaka H, Winter MA, Perkison WB, Brown EL, Aguilar D, Hanis CL. Acculturation, Dietary Behaviors, and Macronutrient Intake Among Mexican Americans With Prediabetes: The Starr County Diabetes Prevention Initiative. Sci Diabetes Self Manag Care. 2023 Feb;49(1):65-76. doi: 10.1177/26350106221146473. Epub 2023 Jan 23. PMID 36683588
- [Derived] Brown SA, Winter MA, Becker HA, Garcia AA, Velasquez MM, Tanaka H, Perkison WB, Brown EL, Aguilar D, Hanis CL. Transitioning From an In-Person Intervention to Augmented Text Messaging During COVID-19 in Mexican Americans With Prediabetes: The Starr County Diabetes Prevention Randomized Clinical Trial. Sci Diabetes Self Manag Care. 2024 Apr;50(2):107-115. doi: 10.1177/26350106241233475. Epub 2024 Mar 7. PMID 38454633

DOCUMENTS (1):
  • Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03208010/ICF_000.pdf